CLINICAL TRIAL: NCT03107338
Title: Effects of the Preoperative Administration of Dexketoprofen Trometamol on Pain and Swelling After Implant Surgery: a Randomized, Double-blind Controlled Trial.
Brief Title: Preventive Treatment of Pain After Dental Implant Surgery
Acronym: UMU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Collaborators: Mozo Grau Ticare (Unknown)
Responsible Party: Principal Investigator, Arturo Sánchez-Pérez, Associate professor, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 30102009
Record Dates: First submitted 2017-03-16; First posted 2017-04-11 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Acute Pain
Keywords: Pre-emptive analgesia; Dexketoprofen trometamol
MeSH Terms: conditions — Acute Pain | interventions — dexketoprofen trometamol

STUDY DESIGN:
Intervention Model Description: This study was conducted as a prospective randomized double-blind study with a placebo. The present study considered the checklist items proposed in the CONSORT statement.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients and the evaluator of the VAS (MMV) were unaware of the results of the randomization and the treatment received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DEXKETOPROFEN TROMETAMOL (Active Comparator): Patients received a dose of 25 mg DKT in an oral suspension 15 minutes before surgery
  Interventions: Drug: DEXKETOPROFEN TROMETAMOL
- Placebo (Placebo Comparator): Patients received a dose of 500 mg Vitamin C in an oral suspension 15 minutes before surgery
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DEXKETOPROFEN TROMETAMOL — Patients who were administered a single dose of 25 mg of DKT 15 minutes before surgery
  Other Names: Enantyum 25
  Arms: DEXKETOPROFEN TROMETAMOL
Other: Placebo — Patients who were administered a single dose of 500 mg of Vitamin C 15 minutes before surgery
  Arms: Placebo

SUMMARY:
The objective of this prospective randomized double-blind study was to evaluate the effects of the preoperative administration of dexketoprofen trometamol (DKT) on the pain perceived by patients after oral surgery for implant placement.

Materials and Method: Single oral doses of 25 mg DKT or PLACEBO were administered 15 minutes before the performance of conventional implant surgery to assess the influence of the DKT on pain as reported by the patients. One hundred patients who required single-implant treatments were randomly distributed into one of the two blinded groups following a preliminary examination. Fifteen minutes before surgery, the patients in the test group were given 25 mg DKT (DKT group), and those in the control group were given 500 mg vitamin C as a placebo (PLACEBO group). The patients' pain intensities were measured using a subjective visual analogue scale of 100 mm in length, and pain was measured over a period of 7 days. Inflammation was assessed using a 5-point Likert scale on days 2 and 7.

DETAILED DESCRIPTION:
A total of 100 consecutive patients (November 2013 to October 2015) scheduled for implant surgery in the University Dental Clinic (Murcia, Spain) were included in this study. All patients were older than 18 and were free of medical and surgical contraindications and systemic disease that would conflict with treatment (American Society of Anesthesiologists (ASA) risk I or II). All participants in the study were able to read, understand and respond to the health questionnaire and were able to sign an informed consent document. This study was performed in accordance with the 2014 revision of the Declaration of Helsinki (General Assembly of the World Medical Association, 2014).

Clinical materials The study protocol was approved by the Ethics Committee of the University of Murcia.

The study was conducted with a double blind randomized design using a visual analogue scale (VAS) of 100 mm to measure pain intensity. The degree of inflammation was measured using a 5-point Likert scale (extremely inflamed, very inflamed, inflamed, somewhat inflamed, and not inflamed).

Patients signed two informed consent forms, one for the implant surgery, and the other for participation in the study; the latter explicitly mentioned the patients' ability to leave the study at any time.

A local anaesthetic composed of lidocaine hydrochloride and epinephrine (20 mg/ml + 0.0125 mg/ml, respectively) was applied (never alveolar nerve block).

All implants had sandblasted and acid-etched surfaces (TiCare Inhex®, Mozo Grau / Ticare, Valladolid, Spain). All implants were placed by the same surgeon (ASP) following the recommendations of the manufacturer (total = 100 implants).

The test group received a dose of 25 mg DKT in an oral suspension 15 minutes before surgery, and the control group received 500 mg vitamin C 15 minutes before surgery. Both solutions were administered in an orange disposable cup to mask the small difference in colour.

ELIGIBILITY:
Inclusion Criteria:

* Good systemic health status (ASA I or II).
* No current pain.
* No use of painkillers in the prior weeks.
* Older than 18 years.
* Oral hygiene index of < 2 (Löe and Silness).
* A minimum of 2 mm of adhered gum.
* A minimum of 8 mm of vertical bone.
* A minimum of 7 mm of vestibule-lingual bone.
* Scheduled to receive a unitary implant.
* Willing to participate in this controlled study.

Exclusion Criteria:

* Pregnant or nursing women.
* The use of any type of medication that might affect the perception of pain.
* Level of pain greater than 40 mm on the VAS before surgery.
* An history of alcohol or drug abuse.
* Requirement for guided regeneration or maxillary sinus lifting procedures.
* Failure to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2015-10-30 (Actual); Study Completion 2015-11-07 (Actual)

PRIMARY OUTCOMES:
Acute pain after implant surgery | 2 years (until complete sample)
  measured by visual analogue scale (VAS) of 100 mm to measure pain intensity

SECONDARY OUTCOMES:
Inflammation | 2 years (until complete sample)
  Degree of inflammation was measured using a 5-point Likert scale (extremely inflamed, very inflamed, inflamed, somewhat inflamed, and not inflamed).

IPD SHARING:
Plan to Share IPD: Yes
All data there will be share by personal e-mail
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Once the results have been published
Access Criteria: Any interested researcher